CLINICAL TRIAL: NCT04239222
Title: Prospective, Feasibility Study to Evaluate Performance, Patient Benefits, and Acceptance of a New Energy Storage and Return Prosthetic Foot
Brief Title: Feasibility Study to Evaluate a New Energy Storage and Return Prosthetic Foot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Otto Bock Healthcare Products GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: OB111
Record Dates: First submitted 2020-01-17; First posted 2020-01-27 (Actual); Results first posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-06

CONDITIONS: Lower Limb Amputation Below Knee (Injury); Lower Limb Amputation Above Knee (Injury); Lower Limb Amputation Knee
Keywords: Prosthetic foot, lower limb amputation
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Randomized cross-over controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Revo-M to Proflex XC (Experimental): Transtibial amputees randomized to start with Revo-M and cross over to Proflex XC
  Interventions: Device: Revo-M; Device: Proflex XC
- Proflex XC to Revo-M (Experimental): Transtibial amputees randomized to start with Proflex XC and cross over to Revo-M
  Interventions: Device: Revo-M; Device: Proflex XC
- Revo-M to Taleo (Experimental): Transfemoral amputees randomized to start with Revo-M and cross over to Taleo
  Interventions: Device: Revo-M; Device: Taleo
- Taleo to Revo-M (Experimental): Transfemoral amputees randomized to start with Taleo and cross over to Revo-M
  Interventions: Device: Revo-M; Device: Taleo

INTERVENTIONS:
Device: Revo-M — Investigational energy storage and return prosthetic foot with using novel elastic elements.
Device: Taleo — Commercially available carbon-fiber energy storage and return foot used as comparative foot for transfemoral amputee subjects
  Arms: Revo-M to Taleo; Taleo to Revo-M
Device: Proflex XC — Commercially available carbon-fiber energy storage and return foot used as comparative foot for transtibial amputee subjects
  Arms: Proflex XC to Revo-M; Revo-M to Proflex XC

SUMMARY:
A prospective, interventional, multicenter pilot study to characterize differences in performance and patient reported outcomes between the Taleo, Proflex XC, and the new Revo prosthetic foot.

DETAILED DESCRIPTION:
The purpose of the Revo-M Study is to characterize differences in performance and patient reported outcomes between the Revo investigational prosthetic foot and a comparative prosthetic foot (Taleo or Proflex XC) when compared to the control foot which is the subject's currently used energy storage and return (ESR) prosthetic foot. The data obtained from this study may also serve to determine the long-term performance of Revo.

ELIGIBILITY:
Inclusion Criteria:

1. Person is 18 years or older.
2. Currently uses an energy storage and return foot.
3. Person has been a unilateral transfemoral (TF), or transtibial (TT) amputee using a prosthesis for at least 1 year.
4. For TF amputees, the person must be wearing an Ottobock Microprocessor-controlled Knee (MPK) with a compatible prosthetic foot
5. Person weighs ≤ 275 lbs (125 kg) size 26-27cm or ≤ 220 lbs (100 kg) size 24-25cm
6. Person is a K3 ambulator based on Medicare Functional Classification Level (MFCL).
7. Prosthetic foot size is 24 to 27 centimeters.
8. Socket Comfort Score of at least 7
9. Ability to read and understand English
10. A person is able and willing to give consent

Exclusion Criteria:

1. Current prosthetic foot is too old or worn out as assessed by the CPO.
2. TT subject with currently fit with a Proflex XC or TF subject currently fit with a Taleo.
3. Patient is pregnant or planning to become pregnant.
4. Person who has a life-threatening medical condition (i.e. terminal cancer, severe heart disease).
5. Person has conditions that would prevent participation and pose increased risk (e.g. unstable cardiovascular conditions that preclude physical activity such as walking, problems with vestibular system, etc.).
6. Ulceration or skin breakdown of the residual limb.
7. Person currently has residual limb issues that significantly reduce their ability to load the prosthesis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-03-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Artificial Limb Specialists, Mesa, Arizona
  - Dankmeyer Prosthetics & Orthotics, Linthicum, Maryland
  - Optimus Prosthetics, Dayton, Ohio
  - Ability P&O, Exton, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD.

REFERENCES:
- [Background] Gallagher P, Franchignoni F, Giordano A, MacLachlan M. Trinity amputation and prosthesis experience scales: a psychometric assessment using classical test theory and rasch analysis. Am J Phys Med Rehabil. 2010 Jun;89(6):487-96. doi: 10.1097/PHM.0b013e3181dd8cf1. PMID 20489393
- [Background] Hafner BJ, Morgan SJ, Askew RL, Salem R. Psychometric evaluation of self-report outcome measures for prosthetic applications. J Rehabil Res Dev. 2016;53(6):797-812. doi: 10.1682/JRRD.2015.12.0228. PMID 28273329

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 Subject failed screening
Period: Baseline
Arm/Group | Revo-M to Proflex XC | Proflex XC to Revo-M | Revo-M to Taleo | Taleo to Revo-M
Started | 6 (The screen failure did not complete baseline assessments) | 8 | 4 | 8
Completed | 6 | 8 | 3 | 7
Not Completed | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1
Period: First Foot Assignment
Arm/Group | Revo-M to Proflex XC | Proflex XC to Revo-M | Revo-M to Taleo | Taleo to Revo-M
Started | 6 | 8 | 3 | 7
Completed | 6 | 8 | 2 | 7
Not Completed | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Period: Crossover to Alternate Foot Assignment
Arm/Group | Revo-M to Proflex XC | Proflex XC to Revo-M | Revo-M to Taleo | Taleo to Revo-M
Started | 6 | 8 | 2 | 7
Completed | 6 | 8 | 1 (One subject could not tolerate the Taleo for any amount of time, and so was not assessed on Taleo) | 7
Not Completed | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Period: Return to Baseline Foot
Arm/Group | Revo-M to Proflex XC | Proflex XC to Revo-M | Revo-M to Taleo | Taleo to Revo-M
Started | 6 | 8 | 2 (Due to the low enrollment in this arm, the subject who could not tolerate Taleo was allowed to finish on the baseline foot) | 7
Completed | 6 | 8 | 2 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Revo-M to Proflex XC | Proflex XC to Revo-M | Revo-M to Taleo | Taleo to Revo-M | Total
Number analyzed (Participants) | 6 | 8 | 4 | 8 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 5 | 4 | 4 | 15
  >=65 years | 4 | 3 | 0 | 4 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (7.9) | 52.4 (16.8) | 44.8 (9.4) | 60.1 (23.5) | 56.3 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 1 | 2 | 5
  Male | 6 | 6 | 3 | 6 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 0 | 1 | 4
  White | 5 | 6 | 4 | 7 | 22
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: centimeters] | 175.0 (4.3) | 170.5 (9.1) | 173.5 (8.7) | 176.1 (61.9) | 173.7 (7.6)
Weight [Mean (Standard Deviation); unit: kilograms] | 88.7 (14.1) | 78.0 (9.8) | 81.8 (7.2) | 92.1 (34.8) | 85.4 (13.4)
Years since amputation [Mean (Standard Deviation); unit: years] | 11.8 (14.9) | 12.6 (14.8) | 22.0 (13.1) | 14.9 (16.3) | 16.2 (15.3)
Amputation level [Count of Participants; unit: Participants]
  Transtibial | 6 | 8 | 0 | 0 | 14
  Transfemoral | 0 | 0 | 4 | 8 | 12
Mobility grade [Count of Participants; unit: Participants] — K1: has ability/potential to use a prosthesis for transfers or ambulation on level surfaces at fixed cadence or speed, typical of a household ambulator.
  K2: has ability/potential for ambulation with the ability to traverse low-level environmental barriers, typical of the limited community ambulator.
  K3: has ability/potential for ambulation with variable cadence or multiple speeds, typically a community ambulator .
  K4: has ability/potential for ambulation that exceeds basic ambulation skills, exhibiting high impact, stress or energy levels, typical of the child, active adult or athlete.
  Participants
    K1 | 0 | 0 | 0 | 0 | 0
    K2 | 0 | 0 | 0 | 0 | 0
    K3 | 6 | 8 | 4 | 8 | 26
    K4 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Patient-perceived Mobility (PLUS-M)™
Description: Perception of mobility as measured by the Prosthetic Limb Users Survey of Mobility (PLUS-M) 12-item short form. The PLUS-M questionnaire provides a T-score that ranges from 21.8 to 71.4. Higher PLUS-M scores correspond with greater mobility. The T-score has a mean of 50 and a standard deviation (SD) of 10. A PLUS-M T-score of 50 represents the mean mobility reported by the development sample. A T-score greater than 57 indicates that the mobility is above the 75th percentile.
Time Frame: baseline, 2 months after fitting with reference foot, Revo-M, or crossover back to baseline foot
Population: ITT analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Baseline: Study assessments with the prosthetic foot used daily by the subject at baseline, prior to using the reference foot or Revo.
- Reference: The reference foot for transtibial amputees was the Pro-Flex XC. The reference foot for transfemoral amputees was the Taleo.
- Revo: The Revo-M version FM 2.0 is an investigational foot, not yet marketed at the time of the study.
  The Revo-M utilizes carbon springs and polyurethane-foam bumpers as elastic elements. These elastic elements allow for a harmonic rollover during stance phase. The proximal connection to other prosthetic components is provided by the aluminum upper part, which contains a pyramid adaptor for this purpose. Furthermore, there is a pivoting joint at the center of the foot within the aluminum upper part that combines with a tension element in the heel region to form a connection to the elastic elements of the foot.
- Final: Study assessments with the prosthetic foot used daily by the subject at baseline, after using the reference foot and Revo.
Arm/Group | Baseline | Reference | Revo | Final
Number analyzed (Participants) | 24 | 22 | 23 | 23
units on a scale | 57.2 (6.6) | 56.9 (7.4) | 58.3 (7.2) | 57.6 (7.1)
Statistical Analysis 1: Comparison: Baseline vs Revo; HO: μRevo-M ≤ μEveryday, μRevo-M is the mean PLUS-M score using the Revo-M and μEveryday is the mean PLUS-M score using the Everyday foot at baseline; Test type: Superiority — A sample size of 22 subjects was required to provide 80% power to detect a difference of 5 points on the PLUS-M scale using Wilcoxon's matched pairs signed ranks test and alpha of 0.05. A standard deviation of 7.7 was used to calculate the sample size; p = 0.286, Wilcoxon Signed Rank Test; Mean Difference (Final Values) = 1.02, Standard Deviation 4.17 — Difference represents Revo-M - Everyday Foot,; 2-sided Wilcoxon matched pairs signed ranks test, n=23 (11 negative, 8 positive and 4 null), Z=-1.066

2. Primary Outcome: Patient-perceived Activity Restrictions (Revised TAPES-AR Subscale)
Description: Activity restrictions as measured by the Revised Trinity Amputation and Prosthesis Experience Scales Activity Restrictions subscale (TAPES-AR). The TAPES-AR subscale has 10 items on a three-point scale and the average score ranges from 0 to 2. A higher score indicates greater activity restriction.
Time Frame: baseline, 2 months after fitting with reference foot, Revo-M, or crossover back to baseline foot
Population: ITT analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline | Reference | Revo | Final
Number analyzed (Participants) | 24 | 22 | 23 | 23
score on a scale | 0.653 (0.362) | 0.686 (0.432) | 0.569 (0.399) | 0.674 (0.388)
Statistical Analysis 1: Comparison: Baseline vs Revo; HO: μRevo-M ≥ μEveryday, μRevo-M is the mean TAPES-AR score using the Revo-M and μEveryday is the mean TAPES-AR score using the Everyday foot at baseline; Test type: Superiority — A sample size of 21 subjects was required to provide 80% power to detect a difference of 0.2 points in the TAPES-AR score using Wilcoxon's matched pairs signed ranks test and alpha of 0.05. A standard deviation of 0.3 was used to calculate the sample size; p = 0.031, Wilcoxon Signed Rank Test; Mean Difference (Final Values) = -0.094, Standard Deviation 0.212 — Difference represents Revo-M - Everyday Foot; 2-sided Wilcoxon matched pairs signed ranks test, n=23 (5 negative, 13 positive and 5 null), Z=-2.156

3. Secondary Outcome: Percentage of Subjects Showing Improvement in Walking Endurance or Perceived Exertion in the 6-minute Walk Test
Description: The percentage of subjects showing an improvement compared to baseline walking endurance as measured by the distance walked in the six minute walk test OR a decrease in the rating of perceived exertion (RPE) as measured by Borg CR100 while wearing the Revo-M. A clinically-significant improvement in the 6MWT is defined as a change in distance of greater than 45 meters. A clinically-significant improvement in the RPE is defined as a change greater than 10 points. The Borg CR100 scale has a minimum of 0 and a maximum of 100. Greater scores indicate higher perceived exertion.
Time Frame: 2 months after fitting with reference foot, Revo-M, or crossover back to baseline foot
Population: ITT analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Reference | Revo | Final
Number analyzed (Participants) | 22 | 23 | 23
Participants | 11 | 8 | 10

4. Secondary Outcome: Patient Perceived Balance Confidence (ABC)
Description: Perception of balance confidence as measured by the extended Activities-specific Balance Confidence (ABC) Scale. The questionnaire provides a score that ranges from 0 to 100%. Higher scores indicate greater balance confidence.
Time Frame: baseline, 2 months after fitting with reference foot, Revo-M, or crossover back to baseline foot
Population: ITT analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline | Reference | Revo | Final
Number analyzed (Participants) | 24 | 22 | 23 | 23
score on a scale | 86.8 (8.9) | 86.2 (11.3) | 87.7 (11.2) | 86.9 (10.9)
Statistical Analysis 1: Comparison: Baseline vs Revo; HO: μRevo-M ≤ μEveryday, μRevo-M is the mean ABC score using the Revo-M and μEveryday is the mean ABC score using the Everyday foot at baseline; Test type: Superiority; p = 0.421, Wilcoxon Signed Rank Test; Mean Difference (Final Values) = 0.331, Standard Deviation 8.29 — Difference represents Revo-M - Everyday Foot; 2-sided Wilcoxon matched pairs signed ranks test, n=23 (12 negative, 7 positive and 4 null), Z=-0.805

5. Secondary Outcome: Functional Satisfaction With Prosthesis (TAPES-FUN)
Description: To characterize the level of functional satisfaction as measured by the TAPES Functional Satisfaction (TAPES-FUN) subscale while wearing a given prosthetic foot. There are 5 items scaled from 1 to 5. The subscale provides a total score that ranges from 5 to 25. Higher scores indicate greater functional satisfaction.
Time Frame: baseline, 2 months after fitting with reference foot, Revo-M, or crossover back to baseline foot
Population: ITT analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline | Reference | Revo | Final
Number analyzed (Participants) | 24 | 22 | 23 | 23
score on a scale | 21.6 (4.3) | 21.5 (3.2) | 22.1 (2.3) | 20.4 (4.6)
Statistical Analysis 1: Comparison: Baseline vs Revo; HO: μRevo-M ≤ μEveryday, μRevo-M is the mean TAPES-FUN score using the Revo-M and μEveryday is the mean TAPES-FUN score using the Everyday foot at baseline; Test type: Superiority; p = 0.443, Wilcoxon Signed Rank Test; Mean Difference (Final Values) = 0.087, Standard Deviation 0.844 — Difference represents Revo-M - Everyday Foot; 2-sided Wilcoxon matched pairs signed ranks test, n=23 (6 negative, 9 positive and 8 null), Z=-0.767

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the four periods in the study. Each home-use period was between 6 to 10 weeks.
Description: For patients with frequent falls or stumbles, an increase in frequency was considered an adverse event and any falls that resulted in an injury were noted individually as adverse events. Seriousness was determined by the consequences of the event as defined in ISO 14155. Due to the expected low rates for adverse events, it was pre-specified to combine adverse events recorded during the Baseline arm with the Everyday Foot with those reported in the Final arm after return to the Everyday Foot.
Groups:
- Everyday Foot: The prosthetic foot used daily by the subject at baseline. Due to the ABCA crossover design, subjects would be expected to spend nearly double the amount of time in this group.
- Reference Foot: The reference foot for transtibial amputees was the Pro-Flex XC. The reference foot for transfemoral amputees was the Taleo.
- Revo-M: The Revo-M version FM 2.0 is an investigational foot, not yet marketed at the time of the study.
  The Revo-M utilizes carbon springs and polyurethane-foam bumpers as elastic elements. These elastic elements allow for a harmonic rollover during stance phase. The proximal connection to other prosthetic components is provided by the aluminum upper part, which contains a pyramid adaptor for this purpose. Furthermore, there is a pivoting joint at the center of the foot within the aluminum upper part that combines with a tension element in the heel region to form a connection to the elastic elements of the foot.
Arm/Group | Everyday Foot | Reference Foot | Revo-M
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/22 | 0/23
Serious Adverse Events (participants affected / at risk) | 1/26 | 1/22 | 2/23
Other Adverse Events (participants affected / at risk) | 3/26 | 7/22 | 6/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Everyday Foot (N=26) | Reference Foot (N=22) | Revo-M (N=23)
Intestinal blockage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bacterial Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Everyday Foot (N=26) | Reference Foot (N=22) | Revo-M (N=23)
Injurious Fall (General disorders) | 0 (0) | 0 (0) | 1 (1)
Bone Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (1)
Muscle Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in hip (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in leg (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral neuropathy aggravated (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Knee Instability (Product Issues) | 0 (0) | 3 (3) | 1 (1) — Only applicable to transfemoral amputees using a prosthetic knee, typically described as the joint feeling "squishy"
Loss of suction (Product Issues) | 0 (0) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Open Wound (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
A small overall sample. One subject could not tolerate the Taleo foot for any amount of time and so was not assessed on the Taleo.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-22): https://cdn.clinicaltrials.gov/large-docs/22/NCT04239222/Prot_SAP_000.pdf